CLINICAL TRIAL: NCT03154827
Title: An Open-Label, Single Arm, Study, To Evaluate the Safety, Tolerability and Efficacy of the BL-8040 and Atezolizumab Combination for Maintenance Treatment in Subjects With Acute Myeloid Leukemia Who Are 60 Years or Older - The BATTLE Study
Brief Title: Safety, Tolerability and Efficacy of the BL-8040 and Atezolizumab for Maintenance Treatment in Subjects With Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to lack of enrollment
Sponsor: BioLineRx, Ltd. (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-8040.AML.202
Record Dates: First submitted 2017-05-14; First posted 2017-05-16 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 4-fluorobenzoyl-TN-14003; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Treatment Single Arm (Experimental): Combination Treatment of BL-8040 with Atezolizumab
  Interventions: Drug: BL-8040; Drug: Atezolizumab

INTERVENTIONS:
Drug: BL-8040 — Subjects will receive maintenance treatment consisting of subcutaneous (SC) injections of BL-8040 on Days 1, 2 and 3 of each 21-day cycle. Cycles will be repeated for up to 2 years (a maximum of 34 treatment cycles), until early discontinuation for any reason or until disease relapse, whichever comes first.
  Other Names: Motixafortide
Drug: Atezolizumab — Subjects will receive maintenance treatment consisting of intravenous (IV) infusion of Atezolizumab on Day 2 of each 21-day cycle. Cycles will be repeated for up to 2 years (a maximum of 34 treatment cycles), until early discontinuation for any reason or until disease relapse, whichever comes first.
  Other Names: Tecentriq

SUMMARY:
A Phase Ib/II, Multicenter, Single Arm, Open-Label Study, To Evaluate the Safety, Tolerability and Efficacy of the BL-8040 and Atezolizumab Combination for Maintenance Treatment in Subjects with Acute Myeloid Leukemia- The BATTLE Study

The main goal of this clinical trial is to assess the safety and tolerability of the treatment combination of BL-8040 and Atezolizumab as Maintenance Treatment in Subjects with Acute Myeloid Leukemia.

Additional objectives are:

Assessment of the effect of combination of BL-8040 and Atezolizumab on relapse free survival (RFS) Assessment whether the treatment combination of BL-8040 and Atezolizumab can reduce the Minimal Residual Disease (MRD) as compared to baseline Assessment of the Overall Survival (OS) time in subjects treated with the combination of BL-8040 and Atezolizumab for maintenance Assessment of the Event Free Survival (EFS) time in subjects treated with the combination of BL-8040 and Atezolizumab for maintenance

DETAILED DESCRIPTION:
This study will assess the safety and effectiveness of a combination of BL-8040 and atezolizumab to find out what is the Safety, Tolerability and Efficacy of this treatment combination for maintenance treatment in subjects with acute myeloid leukemia.

This is a single arm, open label, Phase Ib/II study in which eligible subjects will receive maintenance treatment consisting of intravenous (IV) infusion of Atezolizumab on Day 2 of each 21-day cycle and subcutaneous (SC) injections of BL-8040 on Days 1, 2 and 3 of each 21-day cycle. Cycles will be repeated for up to 2 years (a maximum of 34 treatment cycles), until early discontinuation for any reason or until disease relapse, whichever comes first.

Approximately 60 patients will take part at multiple centers worldwide.

The duration of the treatment period of the study will be up to 2 years and will be followed by one year safety follow up. The study will consist of:

* a screening period of 21 days to allow your doctor to assess your suitability for enrollment into the study
* a treatment period of combination regimen of 21 day cycles for up to 2 years
* a follow-up period of up to 30 days after completion of combined treatment with BL-8040 + Atezolizumab
* an additional follow up period for up to one year after the completion of the treatment

ELIGIBILITY:
Inclusion Criteria:

AML confirmed subjects aged ≥ 60 years who have achieved complete remission (CR or CRi) after induction/consolidation Ara-C based therapy, that have MRD positive status and are not planned for stem cell transplantation.

Exclusion Criteria:

Subjects diagnosed with acute promyelocytic leukemia or with extramedullary AML or subjects who have achieved CR or CRi following treatment for AML. Subjects who have received treatment with hypomethylating agents.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (2):
  - The University of Texas - Md Anderson Cancer Center - Leukemia Center, Houston, Texas
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Czechia (3):
  - Fakultni Nemocnice Brno / University Hospital Brno Interni Hematologicka A Onkologicka Klinika / Internal Hematology and Oncology Clinic, Brno
  - Fakultni Nemocnice Ostrava (Fno) / University Hospital Ostrava Klinika Hematoonkologie / Hematooncology Clinic, Ostrava
  - Fakultni Nemocnice Kralovske Vinohrady Fnkv / University Hospital Kralovske Vinohrady Interní Hematologická Klinika Fnkv / Internal Hematology Clinic, Prague
- Israel (2):
  - Rambam Medical Center, Haifa
  - Shaarei Tzedek Medical Center, Jerusalem
- Wojewódzkie Wielospecjalistyczne Centrum Onkologii I Traumatologii Im. M. Kopernika W Lodzi, Lodz, Poland
- Národný Onkologický Ústav / National Cancer Institute, Oddelenie Onkohematológie Ii / Department of Oncohematology Ii, Bratislava, Slovakia
- Spain (3):
  - Hospital San Pedro de Alcántara de Cáceres, Cáceres
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Treatment Single Arm
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: All patients who were eligible to the study
Groups:
- Combination Treatment of BL-8040 With Atezolizumab: Combination Treatment of BL-8040 with Atezolizumab
  BL-8040: Subjects will receive maintenance treatment consisting of subcutaneous (SC) injections of BL-8040 on Days 1, 2 and 3 of each 21-day cycle. Cycles will be repeated for up to 2 years (a maximum of 34 treatment cycles), until early discontinuation for any reason or until disease relapse, whichever comes first.
  Atezolizumab: Subjects will receive maintenance treatment consisting of intravenous (IV) infusion of Atezolizumab on Day 2 of each 21-day cycle. Cycles will be repeated for up to 2 years (a maximum of 34 treatment cycles), until early discontinuation for any reason or until disease relapse, whichever comes first.
Arm/Group | Combination Treatment of BL-8040 With Atezolizumab
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Czechia | 1

OUTCOME MEASURES:

1. Primary Outcome: Relapse Free Survival
Description: Relapse Free Survival measured from the time of Complete Remission to the relapse or death from any cause whichever comes first
Time Frame: Up to 5 years
Population: All eligible patients who received at least 1 dose of study medications
Arm/Group | Combination Treatment of BL-8040 With Atezolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed from study start upon informed consent signature until end of study which is approximately 1 year
Arm/Group | Combination Treatment of BL-8040 With Atezolizumab
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Treatment of BL-8040 With Atezolizumab (N=1)
Bronchiolitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Treatment of BL-8040 With Atezolizumab (N=1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT03154827/Prot_SAP_000.pdf